CLINICAL TRIAL: NCT00167388
Title: The Effect of Packed Red Blood Cell Transfusion on Superior Mesenteric Artery Blood Flow Velocity in Premature Infants After Feeding
Brief Title: The Effect of Blood Transfusion on Blood Flow to the Intestines of Premature Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Irene McLeneham Young Investigator Award through Magee Womens Research Institute (Unknown)
Responsible Party: Principal Investigator, Toby Yanowitz, Assistant Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0404184
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-04

CONDITIONS: Anemia of Prematurity
Keywords: anemia; prematurity; blood flow velocity; superior mesenteric artery; intestinal blood flow in premature infants
MeSH Terms: conditions — Anemia; Premature Birth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- group 1 (No Intervention): All babies <1250 gm at the time of the study are enrolled into this arm, and randomized to be NPO during the PRBC transfusion
- group 2 (Active Comparator): Babies <1250 gm at the time of the study are enrolled into this arm, and randomized to be fed during the PRBC transfusion
  Interventions: Other: feed during blood transfusion
- group 3 (No Intervention): All babies >1250 gm at the time of the study are enrolled into this arm, and randomized to be fed during the PRBC transfusion
- group 4 (Experimental): All babies <1250 gm at the time of the study are enrolled into this arm, and randomized to be fed during the PRBC transfusion
  Interventions: Other: feed during blood transfusion

INTERVENTIONS:
Other: feed during blood transfusion — babies receiving the intervention are fed during the PRBC transfusion
  Arms: group 2; group 4

SUMMARY:
The purpose of the study is to see if a blood transfusion changes how fast blood flows to the intestines of a premature baby. Blood flow is measured by an ultrasound test. The investigators also look to see if the blood flow to the intestines depends on whether the baby feeds or doesn't feed during the blood transfusion.

DETAILED DESCRIPTION:
Currently a disparity exists among the NICU staff at Magee-Womens Hospital regarding whether premature infants should be fed during a blood transfusion. The effects of a blood transfusion on superior mesenteric artery blood flow velocity and the post-prandial hyperemia are not known.

We hypothesize that the post-prandial change in mesenteric blood flow velocity (BFV) will be the same before as after a packed red blood cell (PRBC) transfusion among anemic premature infants.

Sixty anemic infants (25-32 weeks GA, feeding >= 60 cc/kg/day) will undergo pre- and post-feed superior mesenteric artery Doppler studies both before and after a blood transfusion. Infants will be stratified by current weight into two groups (< 1250 grams and > 1250 grams). In each weight stratum the infants will be randomized to feeding or NPO during the PRBC transfusion. Randomization will be by block design, with block sizes ranging from two to six infants. The investigator performing the Doppler studies will remain masked to the feeding assignment of the infant.

The primary outcome for the study is the superior mesenteric artery blood flow velocity response to feeding between anemic and non-anemic states among premature infants. Our secondary outcome is the effect of feeding on BFV between anemic and non-anemic states in these infants. Statistical analysis will include paired and unpaired Student t-tests and regression analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton infants born at 25-32 weeks gestation who are < 38 weeks post-conceptual age at enrollment
2. First infant of twin gestation born at 25-32 weeks gestation who requires a blood transfusion; if both infants require transfusion on the same day the larger infant will be enrolled.
3. Receiving bolus enteral feeds [PO (bottle) and/or PE (feeding tube)] of at least 60 cc/kg/day
4. A planned packed red blood cell transfusion, as per the clinical team, for anemia
5. Infant is very likely to require a blood transfusion according to the attending neonatologist.

Exclusion Criteria:

1. Known congenital anomalies of the heart, brain, kidneys or intestine
2. Chromosomal abnormality
3. Intrauterine growth restriction at < 3% for weight at birth since this has been shown to alter mesenteric BFV and the post-prandial hyperemia
4. Twin to twin transfusion sequence
5. Higher order multiples
6. Patent ductus arteriosus known to be present or currently being treated
7. History of definite necrotizing enterocolitis Bell Stage 2 or greater
8. Concurrent treatments with antibiotics or steroids
9. Feeding intolerance, defined as gastric aspirate > 30% of feed volume on 3 sequential feeds
10. Concurrent enrollment in another randomized trial
11. Infants discharged or transferred to another facility without having received a PRBC transfusion will be excluded post-hoc.

Ages: 25 Weeks to 38 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2005-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Krimmel, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment is completed
Groups:
- Group 1: <1250 gm at time of study, Fed during PRBC transfusion
- Group 2: <1250 gm at time of study, Not fed during PRBC transfusion
- Group 3: >1250 gm at time of study, Fed during PRBC transfusion
- Group 4: >1250 gm at time of study, Not fed during PRBC transfusion
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 5 | 5 | 6 | 6
Completed Doppler Study | 5 | 5 | 6 | 6
Completed | 5 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Infant born at 25-32 weeks GA at Magee Womens Hospital between October 2005 and November 2007 and received a PRBC transfusion.
  Weight <1250 at time of study and randomized to "feeding" during the PRBC transfusion
- Group 2: Infant born at 25-32 weeks GA at Magee Womens Hospital between October 2005 and November 2007 and received a PRBC transfusion.
  Weight <1250 at time of study and randomized to "not feeding" during the PRBC transfusion
- Group 3: Infant born at 25-32 weeks GA at Magee Womens Hospital between October 2005 and November 2007 and received a PRBC transfusion.
  Weight >1250 at time of study and randomized to "feeding" during the PRBC transfusion
- Group 4: Infant born at 25-32 weeks GA at Magee Womens Hospital between October 2005 and November 2007 and received a PRBC transfusion.
  Weight >1250 at time of study and randomized to "not feeding" during the PRBC transfusion
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 5 | 6 | 6 | 22
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 4 | 15
  Male | 1 | 1 | 3 | 2 | 7
Weight at time of study [Mean (Full Range); unit: grams] | 886 [839 to 1248] | 736 [696 to 1105] | 1752 [1595 to 1945] | 1856 [1409 to 2393] | 1127 [696 to 2393]

OUTCOME MEASURES:

1. Primary Outcome: Change in Superior Mesenteric Artery Blood Flow Velocity From Pre-to-post Feed in the Anemic and the Transfused States
Description: Time-averaged mean and Peak systolic Doppler blood flow velocity in the mesenteric artery was measured before and after a feed when the baby was anemic (pre-PRBC transfusion) and then again when the baby was immediately post-transfusion
Time Frame: 1 hour
Population: the number below represents the change in the parameter with feeding while the baby anemic (pre-transfusion)
Measure: Mean (Standard Deviation); unit: cm/sec
Groups:
- Groups 1 and 2: Infants <1250 gm, irrespective of whether they were fed or NPO during the PRBC transfusion
- Groups 3 and 4: Infants >1250 gm, irrespective of whether they were fed or NPO during the PRBC transfusion
Arm/Group | Groups 1 and 2 | Groups 3 and 4
Number analyzed (Participants) | 10 | 12
cm/sec
  Mean MBFV Response to feeding when anemic | 2.02 (6.15) | 5.91 (4.08)
  Peak Systolic BFV Response to feeds when anemic | 7.66 (14.40) | 14.99 (14.97)
  Mean MBFV Response to Feeding Post-Transfusion | 0.43 (1.91) | 3.61 (2.46)
  Pk Systolic BFV Response to Feed Post-Transfusio | -1.24 (5.53) | 15.24 (6.36)
Statistical Analysis 1: Comparison: Groups 1 and 2; Change in mean mesenteric blood flow velocity from pre- to post- feed in the anemic state for babies <1250 gm; Test type: Superiority or Other; p = 0.571, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Groups 1 and 2; change in peak systolic blood flow velocity from pre-to post feed for babies <1250 gm while anemic; Test type: Superiority or Other; p = 0.345, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Groups 3 and 4; Change in superior mesenteric artery blood flow velocity from pre- to post- feed in the anemic state for babies >1250 gm; Test type: Superiority or Other; p = 0.006, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Groups 3 and 4; change in peak systolic blood flow velocity from pre-to post feed for babies >1250 gm while anemic; Test type: Superiority or Other; p = 0.035, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Groups 1 and 2; Change in mean mesenteric blood flow velocity from pre-to post-feed for babies <1250 gm after the PRBC transfusion; Test type: Superiority or Other; p = 0.910, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Groups 1 and 2; Change in Peak systolic mesenteric blood flow velocity from pre-to post-feed for babies <1250 gm after the PRBC transfusion; Test type: Superiority or Other; p = 0.850, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Groups 3 and 4; Change in mean mesenteric blood flow velocity from pre-to post-feed for babies >1250 gm after the PRBC transfusion; Test type: Superiority or Other; p = 0.507, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Groups 3 and 4; Change in peak systolic mesenteric blood flow velocity from pre-to post-feed for babies >1250 gm after the PRBC transfusion; Test type: Superiority or Other; p = 0.286, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: The main adverse event being evaluated was necrotizing enterocolitis. The did not occur in any infant
Groups:
- Group 1: < 1250 gm Fed during the study
- Group 2: <1250 gm, not fed during the study
- Group 3: >1250 gm, fed during the study
- Group 4: >1250 gm, not fed during the study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes